CLINICAL TRIAL: NCT02570256
Title: Error-enhanced Learning & Recovery in 2 & 3 Dimensions
Brief Title: Deficit Fields for Stroke Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, James Patton, Co-Director, Robotics Laboratory, Sensory Motor Performance Program, Rehabilitation Institute of Chicago, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RehabilitationIC; 2R01NS053606-05A1 (NIH)
Record Dates: First submitted 2015-10-01; First posted 2015-10-07 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2018-10

CONDITIONS: Stroke
Keywords: stroke; upper extremity; motor exploration; error augmentation; robotic rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Deficit-fields to reduce error (Experimental): We hypothesize that a deficit-field design, using the statistics of a patient's errors to customize training, will provide optimal augmentation that varies during motion as needed. We will compare the training effects of error deficit-fields with previous methods of error augmentation to improve reaching ability.
  Interventions: Behavioral: Deficit-fields to reduce error
- Deficit-fields to expand range of motion (Experimental): Amplifying augmentation can expand motor exploration and improve skill retention in patients. Using motor exploration patterns from each patient, we will form customized deficit-fields to recover normal joint workspace. We will compare augmentation training that either amplifies or diminishes the observed deficits (Expt-1). We also compare deficit-fields with our prior augmentation methods to determine the added value of increased customization (Expt-2).
  Interventions: Behavioral: Deficit-fields to expand range of motion
- Deficit-fields to improve function (Experimental): Here we present visual distortion of whole body movement during manual tasks during standing, including reaching, grasping, and object manipulation. We compare the training effects of feedback based on deficit-fields versus practice with normal vision.
  Interventions: Behavioral: Deficit-fields to improve function

INTERVENTIONS:
Behavioral: Deficit-fields to reduce error — Stroke survivors exhibit error in both reaching extent and abnormal curvatures of motion. Prior error augmentation techniques multiply error by a constant at each instant during movement. However, magnification of spurious errors may provoke over-compensation. We hypothesize that a deficit-field design, using the statistics of a patient's errors to customize training, will provide optimal augmentation that varies during motion as needed. We will compare the training effects of error deficit-fields with previous methods of error augmentation to improve reaching ability.
  Arms: Deficit-fields to reduce error
Behavioral: Deficit-fields to expand range of motion — Motor deficits manifest in the workspace limitations of joints, i.e. reduced range of motion, uneven extension-flexion, inter-joint coupling, and unwanted synergies. Our work builds upon these ideas by augmenting self-directed movement for training coordination. We found that amplifying augmentation can expand motor exploration and improve skill retention in patients. Using motor exploration patterns from each patient, we will form customized deficit-fields to recover normal joint workspace. We will compare augmentation training that either amplifies or diminishes the observed deficits (Expt-1). We also compare deficit-fields with our prior augmentation methods to determine the added value of increased customization (Expt-2).
  Arms: Deficit-fields to expand range of motion
Behavioral: Deficit-fields to improve function — Clinicians have recognized the benefits of training on everyday tasks (Hubbard, Parsons et al. 2009), as well as practice with whole-body actions (Boehme 1988; Bohannon 1995). However, typical robotic systems have only a single contact point and cannot drive the multiple joints involved in functional tasks. Visual distortions (e.g. a shift, rotation or stretch) can promote adaptation even without forces. Here we present visual distortion of whole body movement during manual tasks during standing, including reaching, grasping, and object manipulation. We compare the training effects of feedback based on deficit-fields versus practice with normal vision.
  Arms: Deficit-fields to improve function

SUMMARY:
This study investigates the potential of customized robotic and visual feedback interaction to improve recovery of movements in stroke survivors. While therapists widely recognize that customization is critical to recovery, little is understood about how take advantage of statistical analysis tools to aid in the process of designing individualized training. Our approach first creates a model of a person's own unique movement deficits, and then creates a practice environment to correct these problems. Experiments will determine how the deficit-field approach can improve (1) reaching accuracy, (2) range of motion, and (3) activities of daily living. The findings will not only shed light on how to improve therapy for stroke survivors, it will test hypotheses about fundamental processes of practice and learning. This study will help us move closer to our long-term goal of clinically effective treatments using interactive devices.

ELIGIBILITY:
Inclusion Criteria:

STROKE SURVIVORS:

* adult (age >18)
* Chronic stage stroke recovery (8+ months post)
* available medical records and radiographic information about lesion locations
* strokes caused by an ischemic infarct in the middle cerebral artery
* primary motor cortex involvement
* a Fugl-Meyer score (between 15-50) to evaluate arm motor impairment level

HEALTHY CONTROL PARTICIPANTS:

* adult (age >18)
* healthy individuals with no history of stroke or neural injury

Exclusion Criteria:

* bilateral paresis;
* severe sensory deficits in the limb
* severe spasticity (Modified Ashworth of 4) preventing movement
* aphasia, cognitive impairment or affective dysfunction that would influence the ability to perform the experiment
* inability to provide an informed consent
* severe current medical problems
* diffuse/multiple lesion sites or multiple stroke events
* hemispatial neglect or visual field cut that would prevent subjects from seeing the targets.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Arm motor recovery scores on the Fugl-Meyer | Baseline at beginning of week 1 and 3 prior to intervention; post-evaluation at end of week 4; follow-up evaluation at end of week 5
  Change from baseline in arm motor recovery as measured by Fugl-Meyer

SECONDARY OUTCOMES:
Number of blocks transferred in Box and Blocks Test | Baseline at beginning of week 1 and 3 prior to intervention; post-evaluation at end of week 4; follow-up evaluation at end of week 5
  Change from baseline in number of blocks transferred during Box and Blocks Test
Modified Ashworth Scale (MAS) | Baseline at beginning of week 1 and 3 prior to intervention; post-evaluation at end of week 4; follow-up evaluation at end of week 5
  Change from baseline in amount of spasticity in elbow flexors and extensors
Elbow active range of motion (ROM) | Baseline at beginning of week 1 and 3 prior to intervention; post-evaluation at end of week 4; follow-up evaluation at end of week 5
  Change from baseline measured in degrees for elbow flexion and extension
Chedoke McMaster Stroke Assessment for Hand | Baseline at beginning of week 1 and 3 prior to intervention; post-evaluation at end of week 4; follow-up evaluation at end of week 5
  Change in baseline in amount of hand motor recovery as measured by Chedoke scale
Time and completion score for Action Research Arm Test (ARAT) | Baseline at beginning of week 1 and 3 prior to intervention; post-evaluation at end of week 4; follow-up evaluation at end of week 5
  Change in baseline score and time for completion of functional measures as part of ARAT

CONTACTS AND LOCATIONS:
Overall Officials: James L Patton, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Wright ZA, Majeed YA, Patton JL, Huang FC. Key components of mechanical work predict outcomes in robotic stroke therapy. J Neuroeng Rehabil. 2020 Apr 21;17(1):53. doi: 10.1186/s12984-020-00672-8. PMID 32316977